CLINICAL TRIAL: NCT05469945
Title: Lower Limb Lymphedema After Gyneco-oncologic Therapy: Can we Prevent Irreversible Lymphedema?
Brief Title: Lymphedema After Gyneco-oncologic Treatment
Acronym: Gynolymph
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Hospital, Louvain (Unknown); Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC 09915
Record Dates: First submitted 2021-09-06; First posted 2022-07-22 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Lymphedema; Genital Neoplasm
Keywords: Lymphedema of the lower limb; Gynaecologic cancer; Sexual well-being; Quality of Life; Cost-investment; Time-investment
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial evaluating the added value of CC2 compressive garments in stage 0-1 LLL
Masking Description: No masking possible: the patient and the provider are well aware of yes or no wearing of compressive garments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm: no compressive garments (No Intervention): Patients detected with early stage LLL (0-1 ISL stadia) start with education and preventive measures.
- Interventional arm: start of CC2 compressive garments (Experimental): Patients in the experimental arm and detected with early stage LLL (0-1 ISL stadia) start with CC2 compressive garments in addition to education and preventive measures.
  Interventions: Device: Compressive garments class II

INTERVENTIONS:
Device: Compressive garments class II — Daily wearing of compressive garments, especially during prolonged standing upright or strenuous activities.
  Other Names: Flat knit Medi Cosy compression class II stockings and/or bermuda
  Arms: Interventional arm: start of CC2 compressive garments

SUMMARY:
Trial developed to inventory the incidence of early and advanced stage lower limb lymphedema in patients diagnosed with and treated for gynaecologic cancer.

Four hundred patients with diagnosis stage 1-3 gynaecologic cancer will be included in an observational cohort between diagnosis until maximum 2 weeks after start of the first treatment. They will be followed for occurrence of lower limb lymphedema up till 2 years after their last treatment.

Data on signs and symptoms, quality of life, time investment and financial expenses will be collected, to provide information on the incidence and risk factors for lower limb lymphedema, and on its impact on patients, regarding quality of life, sexual well-being and time- and financial investment.

Patients developing early stage LLL enter an interventional sub-cohort, in which the effect of class II compressive garments on preventing evolution towards advanced stage LLL will be evaluated.

DETAILED DESCRIPTION:
Context of the problem: Improved knowledge on the diagnosis and treatment of cancer has resulted in an increased number of cancer survivors. Consequently, more patients are confronted, often life-long, with the complications of their cancer treatment. These chronic conditions impact daily functioning and quality of life (QoL), complicate the return to work and undermine psycho-social well-being. One of the most frequent and disabling complications is lymphedema, a condition undermining QoL to an extent exceeding even a 10-year age increase.

The damage of lymphedema covers many aspects of daily life: it changes body image and complicates daily activities as basic as clothing, it increases patient-related health expenditures for treatment and for coping with the disease, reduces patient autonomy in daily functioning and can even cause sensory or motor dysfunctions. So far, no definitive cure exists for lymphedema: patients are confined to life-long preventive measures, compression therapy and regular manual lymph drainage. Surgical repair may be an option in selected cases, but evidence on surgical techniques is limited and their long-term effects are still unknown. Moreover, even after successful repair, conservative treatment is still needed.

Most studies on lymphedema are limited to upper limb lymphedema (ULL), mainly after breast cancer treatment. Only a few publications focus on lower limb lymphedema (LLL), despite its detrimental impact on QoL. This could be due to the difficulties to diagnose and treat LLL in comparison to ULL: LLL often occurs bilaterally or at the level of the groins or genital region, hence impeding diagnosis through comparison. Perimetric measurement of large cone-like oedematous legs is cumbersome. Manual lymph drainage and application of compressive garments is more strenuous for legs than for arms, and the typical bilateral occurrence and large volumes of LLL inflate the cost of treatment garments. However limited, some groups did evaluate the incidence of LLL after pelvic treatment, but maintained the criteria for advanced stage lymphedema as cut off, thereby underestimating the prior phases in which patients are confronted with functional impairment due to LLL, without apparent swelling.

The observational cohort in this study is aimed at inventorying the incidence, timing and risk factors of early as well as advanced stage lymphedema. Time and cost-investment of patients for prevention and/or treatment of LLL will be analyzed. The impact of LLL on QoL and on sexual well-being will be calculated.

A sub-cohort of this trial is of interventional design: in patients, included in the observational cohort and developing early stage LLL, standard of care treatment will be started, including skin care, active exercises and manual lymph drainage. In the experimental group, compressive garments class II will be added and compliance as well as tolerance of these garments will be analyzed.

Side-kicks of this trial are the standardization of perimetric measurements of the legs, validation of a self-report LLL screening tool and testing of the sensitivity and specificity of ICG fluoroscopy to detect early stage LLL.

Sample size calculation:

The sample size is calculated for the interventional sub-cohort, to have at least 80% power to detect a difference between the compression group and the control group for progression of lymphedema. An alpha has been set equal to 0.05.

Sample size calculation is based on evaluation at year 1. No longitudinal analysis is foreseen as primary analysis, but this could be included as a secondary analysis using a GEE analysis.

To detect a difference, in the interventional sub-cohort 109 subjects are required per group (2*109=218 subjects in total for the two groups) to have at least 80% power. If 66% of the patients in the observational cohort will meet the inclusion criteria for the interventional randomized trial, at least 330 (=218/0.66) patients should be included in the observational cohort. To correct for drop out we planned to include 400 patients. This number is feasible within the planned recruitment period of 18-24 months. If the number of subjects would be reached before the end of the planned recruitment period, recruitment will be stopped at 400 patients. If the number is not attained, the recruitment period will be prolonged. If the number of 218 subjects is reached in the interventional sub-cohort, randomization will be stopped and analysis starts. However, the observational cohort will continue accrual until 400 subjects are reached.

We assume a difference in true transition rates (T1 to T3) in both study arms, with 0.4 in the interventional group versus 0.75 in the control group. The recruitment of 109 patients in each treatment arm would allow the assessment of benefit of the intervention with 80% power, based on the 95% two-sided confidence interval approach for the differences in two independent proportions.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (ICF)
* Female patient, recently diagnosed with gynaecologic cancer (cervix, endometrium, vulva, vagina, ovaries…) and candidate for curative treatment
* Age ≥ 18 years
* Understanding of the Dutch language
* Able to understand the informed consent and willing to comply with the protocol, including use of diary or app and timely completion of requested questionnaires.

Exclusion Criteria:

* History of treatment for gynaecologic cancer
* Concurrent second primary tumor(s)
* Pregnancy or pregnancy planned within 2 years
* Known metastasized cancer at the time of inclusion (D0)
* Severe injury, surgery or deformation of the legs or groins in the past
* Vascular malformation of the leg or untreated venous insufficiency with oedema (CEAP C4 or more)
* Mental or psychological problems, inability to comply to the study protocol
* First treatment administered > 2 weeks before
* Clinical signs and symptoms of lymphedema present (ISL stage 0 or higher) at the moment of intake

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of LLL | From diagnosis until 2 years after last oncologic treatment
  Number of patients with transition (evolution) to stage 0-3 LLL (ISL criteria) in the first two years after treatment for gynecologic cancer.
  We defined three potential transitions:
  * T1: from no LLL to reversible stage 0-1 LLL
  * T2: from no LLL to irreversible stage 2-3 LLL
  * T3: from stage 0-1 LLL to stage 2-3 LLL
Incidence rate of transition from stage 0-1 LLL to stage 2-3 LLL in randomized subgroup | From transition to stage 0-1 LLL until 1 year after
  Number of patients diagnosed with stage 0-1 LLL within one year after treatment for gynecologic cancer and that evolve from stage 0-1 LLL to stage 2-3 LLL

SECONDARY OUTCOMES:
Timing of development of LLL | From diagnosis until 2 years after last oncologic treatment
  Registration of the timing of development of the different stages of LLL within the first two years after end of treatment
Risk factors for developing LLL - per age category the number of patients that develop lower limb lymph-edema as assessed with ISL criteria | From diagnosis until 2 years after last oncologic treatment
  Age: the amount of time something has been alive or has existed (years)
Risk factors for developing LLL - weight | From diagnosis until 2 years after last oncologic treatment
  Weight: In the operational definition, the weight of an object is the force measured by the operation of weighing it, which is the force it exerts on its support, expressed in kilograms (kg)
Risk factors for developing LLL - height | From diagnosis until 2 years after last oncologic treatment
  Height: measure of vertical extent (how "tall" something or someone is) (expressed in meters)
Risk factors for developing LLL - per BMI category the number of patients that develop lower limb lymph-edema as assessed with ISL criteria (reported value) | From diagnosis until 2 years after last oncologic treatment
  Body mass index (BMI) is a value derived from the mass (weight) and height of a person. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
Risk factors for developing LLL - per category of physical activity the number of patients that develop lower limb lymph-edema as assessed with ISL criteria | From diagnosis until 2 years after last oncologic treatment
  Physical activity is defined as any voluntary bodily movement produced by skeletal muscles that requires energy expenditure. Physical activity encompasses all activities, at any intensity, performed during any time of day or night. It includes both exercise and incidental activity integrated into daily routine. This integrated activity may not be planned, structured, repetitive or purposeful for the improvement of fitness, and may include activities such as walking to the local shop, cleaning, working, active transport etc.
  Expressed in intensity level (categorical)
Risk factors for developing LLL - Marital status | From diagnosis until 2 years after last oncologic treatment
  Civil status, or marital status, are the distinct options that describe a person's relationship with a significant other. Married, single, divorced, and widowed are examples of civil status.
  Expressed in definition (categorical - married, divorced, widowed, single...)
Risk factors for developing LLL - obstetrical status | From diagnosis until 2 years after last oncologic treatment
  Obstetrical history: medical specialty dealing with the care of all women's reproductive tracts and their children during pregnancy (prenatal period), childbirth and the postnatal period Obstetric state: gravida - partus - abortus - mater
Risk factors for developing LLL - education status | From diagnosis until 2 years after last oncologic treatment
  The International Standard Classification of Education (ISCED 2011) is a statistical framework for organizing information on education maintained by the United Nations Educational, Scientific and Cultural Organization (UNESCO). It is a member of the international family of economic and social classifications of the United Nations.
  Categorical: lower secondary education, upper secondary education, Bachelor's or equivalent, Master's or equivalent, Doctorate or equivalent...
Risk factors for developing LLL - employment status | From diagnosis until 2 years after last oncologic treatment
  Work or labor (or labour in British English) is intentional activity people perform to support themselves, others, or the needs and wants of a wider community Categorical: unemployed, employee, self-employed, retired, student, work-incapacity...
Risk factors for developing LLL - smoking status | From diagnosis until 2 years after last oncologic treatment
  Smoking is a practice in which a substance is burned and the resulting smoke is typically breathed in to be tasted and absorbed into the bloodstream.
  Expressed in categories (never, used to smoke, active smoker)
Risk factors for developing LLL - pack-years | From diagnosis until 2 years after last oncologic treatment
  Smoking is a practice in which a substance is burned and the resulting smoke is typically breathed in to be tasted and absorbed into the bloodstream.
  A pack-year is a clinical quantification of cigarette smoking used to measure a person's exposure to tobacco. This is used to assess their risk of developing lung cancer or other pathologies related to tobacco use.
  Calculation: Number of pack-years = (number of cigarettes smoked per day/20) × number of years smoked. (1 pack has 20 cigarettes in some countries)
Risk factors for developing LLL - alcohol intake | From diagnosis until 2 years after last oncologic treatment
  An alcoholic drink (also called an alcoholic beverage, adult beverage, or simply a drink) is a drink that contains ethanol, a type of alcohol produced by fermentation of grains, fruits, or other sources of sugar that acts as a drug.
  Expressed in categories: never, occasionally, daily
Risk factors for developing LLL - physical appearance | From diagnosis until 2 years after last oncologic treatment
  Human physical appearance is the outward phenotype or look of human beings. Registered as importance adhered to physical appearance on a rating scale from 1 to 10.
  Expressed on a scale of one to ten, (this scale is a general and largely vernacular concept used for rating things, people, places, ideas, and so on. The scale has 10 as a maximum score, as a denotation of exceptionally high quality or of another attribute, a minimum of 0.)
Risk factors for developing LLL - household income category | From diagnosis until 2 years after last oncologic treatment
  Household income is an economic standard that can be applied to one household, or aggregated across a large group such as a county, city, or the whole country. It is commonly used by government and private institutions to describe a household's economic status or to track economic trends.
  Expressed in categories (per month): <1500, 1500-3000, >3000-5000, >5000 or 'does not wish to respond'
Risk factors for developing LLL - number of patients with contact allergy that develop lower limb lymph-edema as assessed with ISL criteria | From diagnosis until 2 years after last oncologic treatment
  Allergies, also known as allergic diseases, are a number of conditions caused by hypersensitivity of the immune system to typically harmless substances in the environment.
Risk factors for developing LLL - number of patients with medical record of disease (renal, cardiac, diabetic...) that develop lower limb lymph-edema as assessed with ISL criteria | From diagnosis until 2 years after last oncologic treatment
  The medical history, case history, or anamnesis of a patient is information gained by a physician by asking specific questions, with the aim of obtaining information useful in formulating a diagnosis and providing medical care to the patient.
  Expressed in relevant categories (cardiac, renal, vascular, cancer, auto-immune...)
Risk factors for developing LLL - pain score | From diagnosis until 2 years after last oncologic treatment
  A pain scale measures a patient's pain intensity or other features. Pain scales are a common communication tool in medical contexts, and are used in a variety of medical settings.
  Expressed on a scale of one to ten, (this scale is a general and largely vernacular concept used for rating things, people, places, ideas, and so on. The scale has 10 as a denotation of exceptionally high pain, and a minimum of 0 for no pain at all.)
Risk factors for developing LLL - tumor stage (TNM) | From diagnosis until 2 years after last oncologic treatment
  The TNM Classification of Malignant Tumors (TNM) is a globally recognised standard for classifying the extent of spread of cancer. It is a classification system of the anatomical extent of tumor cancers.
  Most common tumors have their own TNM classification. Sometimes also described as the AJCC system.
  TNM is a notation system that describes the stage of a cancer, which originates from a solid tumor, using alphanumeric codes:
  T describes the size of the original (primary) tumor and whether it has invaded nearby tissue, N describes nearby (regional) lymph nodes that are involved, M describes distant metastasis (spread of cancer from one part of the body to another).
Risk factors for developing LLL - tumor stage (FIGO) | From diagnosis until 2 years after last oncologic treatment
  The International Federation of Gynaecology and Obstetrics, usually just FIGO as the acronym of its French name Fédération Internationale de Gynécologie et d'Obstétrique, is a worldwide non-governmental organisation representing obstetricians and gynaecologists in over one hundred territories.
  The FIGO staging system is used most often for cancers of the female reproductive organs, including cervical cancer, endometrial cancer, ovarian cancer...
  As a rule, the lower the number, the less the cancer has spread. A higher number, such as stage IV, means a more advanced cancer. And within a stage, an earlier letter means a lower stage. Cancers with similar stages tend to have a similar outlook and are often treated in much the same way.
Risk factors for developing LLL - the number of patients with limited (only one or two gynaecologic organs) or extensive surgery (multiple organs and/or lymph nodes) that develop lower limb lymph-edema as assessed with ISL criteria | From diagnosis until 2 years after last oncologic treatment
  Gynecological surgery refers to surgery on the female reproductive system usually performed by gynecologists. In the domain of cancer it may include hysterectomy, ovariectomy, pelvic exenteration, salpingoophorectomy, vulvectomy and partial or complete lymphadenectomy
Risk factors for developing LLL - the number of patients receiving systemic therapy that develop lower limb lymph-edema as assessed with ISL criteria | From diagnosis until 2 years after last oncologic treatment
  Systemic therapy is a therapy that is given in addition to the primary or initial therapy to maximize its effectiveness. It can be given in adjuvant or neo-adjuvant setting.
  Categorical: none, taxanes, cisplatinum, immunotherapy, target therapy, anti-hormone therapy, other.
Risk factors for developing LLL - the number of patients receiving radiotherapy that develop lower limb lymph-edema as assessed with ISL criteria | From diagnosis until 2 years after last oncologic treatment
  Radiation therapy or radiotherapy, often abbreviated RT, RTx, or XRT, is a therapy using ionizing radiation, generally provided as part of cancer treatment to control or kill malignant cells and normally delivered by a linear accelerator. Radiation therapy may be curative in a number of types of cancer if they are localized to one area of the body. It may also be used as part of adjuvant therapy, to prevent tumor recurrence after surgery to remove a primary malignant tumor (for example, early stages of breast cancer). Radiation therapy is synergistic with chemotherapy, and has been used before, during, and after chemotherapy in susceptible cancers.
  Expressed per target volume in dose per fraction, number of fractions
Impact of LLL on QoL - EQ5D | From diagnosis until 2 years after last oncologic treatment
  EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys. EQ-5D assesses health status in terms of five dimensions of health and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition. EQ-5D can also be referred to as a patient-reported outcome (PRO) measure, because patients can complete the questionnaire themselves to provide information about their current health status and how this changes over time. 'EQ-5D' is not an abbreviation and is the correct term to use when referring to the instrument in general.
  Expressed as an overall measure of self-assessed health status (EQ VAS) at different time points (D0, M3, M12)
Impact of LLL on QoL - EORT qlq C30 | From diagnosis until 2 years after last oncologic treatment
  European Organisation for Research and Treatment of Cancer (EORTC): qlq C30: questionnaire developed by the EORTC and validated in over 100 languages, in order to assess in 30 questions the quality of life of cancer patients.
Impact of LLL on QoL - lymph-ICF-LL | From diagnosis until 2 years after last oncologic treatment
  Lymphoedema Functioning, Disability and Health Questionnaire for Lower Limb Lymphoedema (Lymph-ICF-LL): it is a descriptive, evaluative tool containing 28 questions about impairments in function, activity limitations, and participation restrictions in patients with lower limb lymphedema. The questionnaire has 5 domains: physical function, mental function, general tasks/household activities, mobility activities, and life domains/social life.
Impact of LLL on sexuality | From diagnosis until 2 years after last oncologic treatment
  Female Sexual Distress Scale Revised (FSDS-R) is a multi-dimensional self-reporting questionnaire containing 13 items to evaluate sexual distress in women.
  Evaluation: Percentage of patients with clinically relevant loss in sexual well-being, measured through questionnaire at baseline, 3 months, 12 months and 24 months post-treatment
Predictive value of the self-report LLL questionnaire | From diagnosis until 2 years after last oncologic treatment
  The self-report lower-extremity lymphedema screening questionnaire is a screening questionnaire developed to detect lower-extremity lymphedema (LEL) among normal-weight women and women with obesity.
  Evaluation: Number of patients with score >5 on the self-report LLL questionnaire that are diagnosed with LLL according to ISL criteria (positive predictive value)
Value of ICG fluoroscopy versus lymphoscintigraphy in detection of early stage LLL | From diagnosis until 2 years after last oncologic treatment
  Percentage of positive ICG fluoroscopy (image of splash, stardust or diffuse ICG pattern) corresponding with positive lympho-scintigraphy (signs of impaired lymphatic flow) or with clinical diagnosis of LLL based on ISL criteria
Inventory of time investment | From diagnosis until 2 years after last oncologic treatment
  Calculation of mean time investment of patients in the prevention and treatment of LLL through app-based registration
Inventory of expenses | From diagnosis until 2 years after last oncologic treatment
  Calculation of mean financial investment of patients in the prevention and treatment of LLL through app-based registration
Standardization of perimetric measurements | From diagnosis until 2 years after last oncologic treatment
  Development of standardized instructions for perimetric measurement with measurement from a fixed start point and then every 4cm to calculate leg circumference. Verification of reliability through intra- and interobserver comparison

OTHER OUTCOMES:
Tolerance of and compliance to preventive compressive garments as assessed with the ICC compression questionnaire | From transition to stage until 1 year after
  Satisfaction with compressive garments assessed with ICC compression questionnaire, evaluation of functioning, symptoms of LLL, side-effects of compressive garments, feasibility of use, frequency and duration of wearing, autonomy, improvement or deterioration of functioning on social and job-level
Impact of preventive compressive garments on evolution of leg volume | From transition to stage until 1 year after
  Comparison of evolution of leg circumference measurement between the intervention group (compressive garments and the control group (no compressive garments), measuring leg circumference every 4cm, starting from a fixed point above the ankles to 17 measuring points above. Estimation of volume per leg is based on the truncated cone formula.
Impact of preventive compressive garments on patient's time investment, including putting on and of compressive garments, washing compressive clothing, skin care... | From transition to stage until 1 year after
  Inventory of mean time-investment of patients in the treatment of LLL through app-based registration, and comparison of time-investment between control group (no compressive garments) and interventional group (with compressive garments)
Impact of preventive compressive garments on financial investment, including reimbursed as well as out-of-pocket patient cost for compressive stockings, supplementary tools, nursing aid... | From transition to stage until 1 year after
  Inventory of mean financial investment of patients in the treatment of LLL through app-based registration, and comparison of time-investment between control group (no compressive garments) and interventional group (with compressive garments)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Monten, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Dept. Radiotherapy-Oncology, Ghent
  - University Hospital, Louvain, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yost KJ, Cheville AL, Weaver AL, Al Hilli M, Dowdy SC. Development and validation of a self-report lower-extremity lymphedema screening questionnaire in women. Phys Ther. 2013 May;93(5):694-703. doi: 10.2522/ptj.20120088. Epub 2013 Jan 3. PMID 23288911
- [Background] Hareyama H, Hada K, Goto K, Watanabe S, Hakoyama M, Oku K, Hayakashi Y, Hirayama E, Okuyama K. Prevalence, classification, and risk factors for postoperative lower extremity lymphedema in women with gynecologic malignancies: a retrospective study. Int J Gynecol Cancer. 2015 May;25(4):751-7. doi: 10.1097/IGC.0000000000000405. PMID 25723779
- [Background] Mendivil AA, Rettenmaier MA, Abaid LN, Brown JV 3rd, Micha JP, Lopez KL, Goldstein BH. Lower-extremity lymphedema following management for endometrial and cervical cancer. Surg Oncol. 2016 Sep;25(3):200-4. doi: 10.1016/j.suronc.2016.05.015. Epub 2016 May 20. PMID 27566023
- [Background] Biglia N, Zanfagnin V, Daniele A, Robba E, Bounous VE. Lower Body Lymphedema in Patients with Gynecologic Cancer. Anticancer Res. 2017 Aug;37(8):4005-4015. doi: 10.21873/anticanres.11785. PMID 28739682
- [Background] Carlson JW, Kauderer J, Hutson A, Carter J, Armer J, Lockwood S, Nolte S, Stewart BR, Wenzel L, Walker J, Fleury A, Bonebrake A, Soper J, Mathews C, Zivanovic O, Richards WE, Tan A, Alberts DS, Barakat RR. GOG 244-The lymphedema and gynecologic cancer (LEG) study: Incidence and risk factors in newly diagnosed patients. Gynecol Oncol. 2020 Feb;156(2):467-474. doi: 10.1016/j.ygyno.2019.10.009. Epub 2019 Dec 16. PMID 31837831
- [Background] De Vrieze T, Gebruers N, Nevelsteen I, De Groef A, Tjalma WAA, Thomis S, Dams L, Van der Gucht E, Penen F, Devoogdt N. Reliability of the MoistureMeterD Compact Device and the Pitting Test to Evaluate Local Tissue Water in Subjects with Breast Cancer-Related Lymphedema. Lymphat Res Biol. 2020 Apr;18(2):116-128. doi: 10.1089/lrb.2019.0013. Epub 2019 Jul 19. PMID 31329510
- [Background] Dean LT, Moss SL, Ransome Y, Frasso-Jaramillo L, Zhang Y, Visvanathan K, Nicholas LH, Schmitz KH. "It still affects our economic situation": long-term economic burden of breast cancer and lymphedema. Support Care Cancer. 2019 May;27(5):1697-1708. doi: 10.1007/s00520-018-4418-4. Epub 2018 Aug 18. PMID 30121786
- [Background] Finnane A, Hayes SC, Obermair A, Janda M. Quality of life of women with lower-limb lymphedema following gynecological cancer. Expert Rev Pharmacoecon Outcomes Res. 2011 Jun;11(3):287-97. doi: 10.1586/erp.11.30. PMID 21671698
- [Background] Executive Committee. The Diagnosis and Treatment of Peripheral Lymphedema: 2016 Consensus Document of the International Society of Lymphology. Lymphology. 2016 Dec;49(4):170-84. PMID 29908550
- [Background] Roberson ML, Strassle PD, Fasehun LO, Erim DO, Deune EG, Ogunleye AA. Financial Burden of Lymphedema Hospitalizations in the United States. JAMA Oncol. 2021 Apr 1;7(4):630-632. doi: 10.1001/jamaoncol.2020.7891. PMID 33599683
- [Background] Lindqvist E, Wedin M, Fredrikson M, Kjolhede P. Lymphedema after treatment for endometrial cancer - A review of prevalence and risk factors. Eur J Obstet Gynecol Reprod Biol. 2017 Apr;211:112-121. doi: 10.1016/j.ejogrb.2017.02.021. Epub 2017 Feb 22. PMID 28242470
- [Background] Rockson SG, Rivera KK. Estimating the population burden of lymphedema. Ann N Y Acad Sci. 2008;1131:147-54. doi: 10.1196/annals.1413.014. PMID 18519968
- [Background] Devoogdt N, De Groef A, Hendrickx A, Damstra R, Christiaansen A, Geraerts I, Vervloesem N, Vergote I, Van Kampen M. Lymphoedema Functioning, Disability and Health Questionnaire for Lower Limb Lymphoedema (Lymph-ICF-LL): reliability and validity. Phys Ther. 2014 May;94(5):705-21. doi: 10.2522/ptj.20130285. Epub 2014 Jan 10. PMID 24415775
- [Background] Rowlands IJ, Beesley VL, Janda M, Hayes SC, Obermair A, Quinn MA, Brand A, Leung Y, McQuire L, Webb PM; Australian National Endometrial Cancer Study Group. Quality of life of women with lower limb swelling or lymphedema 3-5 years following endometrial cancer. Gynecol Oncol. 2014 May;133(2):314-8. doi: 10.1016/j.ygyno.2014.03.003. Epub 2014 Mar 11. PMID 24631452
- [Background] Sawan S, Mugnai R, Lopes Ade B, Hughes A, Edmondson RJ. Lower-limb lymphedema and vulval cancer: feasibility of prophylactic compression garments and validation of leg volume measurement. Int J Gynecol Cancer. 2009 Dec;19(9):1649-54. doi: 10.1111/IGC.0b013e3181a8446a. PMID 19955953
- [Background] Stuiver MM, de Rooij JD, Lucas C, Nieweg OE, Horenblas S, van Geel AN, van Beurden M, Aaronson NK. No evidence of benefit from class-II compression stockings in the prevention of lower-limb lymphedema after inguinal lymph node dissection: results of a randomized controlled trial. Lymphology. 2013 Sep;46(3):120-31. PMID 24645535
- [Background] Tartaglione G, Pagan M, Morese R, Cappellini GA, Zappala AR, Sebastiani C, Paone G, Bernabucci V, Bartoletti R, Marchetti P, Marzola MC, Naji M, Rubello D. Intradermal lymphoscintigraphy at rest and after exercise: a new technique for the functional assessment of the lymphatic system in patients with lymphoedema. Nucl Med Commun. 2010 Jun;31(6):547-51. doi: 10.1097/MNM.0b013e328338277d. PMID 20215978
- [Derived] Decorte T, Van Besien V, Van Calster C, Vanden Bossche L, Randon C, Devoogdt N, Monten C. Addition of prophylactic compression garments to standard care to prevent irreversible lower limb lymphoedema after gynaeco-oncological therapy (Gynolymph): protocol for a randomised controlled trial embedded within an observation cohort study. BMJ Open. 2024 Nov 1;14(10):e088851. doi: 10.1136/bmjopen-2024-088851. PMID 39486824